CLINICAL TRIAL: NCT04357743
Title: Effects of Pursed Lip Breathing With Arm Ergometry After Chin Supported Position in COPD Patients.
Brief Title: Pursed Lip Breathing With Arm Ergometry After Chin Supported Position in COPD Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00591 Mashaal Rana
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: COPD
Keywords: Arm Ergometry; Chin Support Position; Oxygen Saturation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chin supported Arm ergometry with pursed lip breathing (Experimental): Chin supported along with Arm ergometry with pursed lip breathing
  Interventions: Other: Chin supported Arm ergometry with pursed lip breathing
- Arm ergometry with pursed lip breathing (Active Comparator): Arm ergometry with pursed lip breathing
  Interventions: Other: Arm ergometry with pursed lip breathing

INTERVENTIONS:
Other: Chin supported Arm ergometry with pursed lip breathing — The participants sat in chin support position for 10 minutes followed by arm ergometry with pursed lip breathing for 10 minutes. The participants again sat in chin support position for 10 minutes.
  The treatment was provided for one week
  Arms: Chin supported Arm ergometry with pursed lip breathing
Other: Arm ergometry with pursed lip breathing — The participants sat in normal position for 10 minutes followed by arm ergometry with pursed lip breathing for 10 minutes; the participants again sat in sitting position for 10 minutes.
  The treatment was provided for one week.
  Arms: Arm ergometry with pursed lip breathing

SUMMARY:
Randomized control Trial, Purposive sampling was used to obtain the sample for the study and then randomly allocated into groups by coin toss method. Data collected from July 2019 to January 2020, was conducted at Rehman Medical Institute Peshawar. To determine the effects of pursed lip breathing with arm ergometry after chin support position on heart rate, respiratory parameters, pulmonary function tests and quality of life in COPD patients.

DETAILED DESCRIPTION:
Chronic Obstructive Lung Disease (COPD), a major worldwide epidemic is the 4th leading cause of death around the globe and though, with rise in worldwide life expectancy and tobacco smoking, predominantly in developing countries, it is likely to be the 3rd leading cause of mortality by 2020. In Pakistan, mortality rate caused by COPD is expected to reach 71 deaths per 100,000 that is globally the fourth leading death rate among 25 most populated countries.

The condition is in the focus worldwide, since its increased prevalence, morbidity and mortality rate create alarming challenges for health-care professionals. In spite of latest trends in decline of COPD consistent death rates and few current achievements in anti-smoking efforts in many western countries, the elevating influence of increasing age in an ever-growing global population, combined with factors as high smoking rates and pollution of air in Asia, will confirm that COPD will last as an ever-increasing issue into the 21st century.

A variety of environmental and intrinsic risk factors are involved in the development of COPD which affect at different time points during an individual's life span. Smoking is a dominant risk factor comprising of 80% of the COPD cases.

During the previous 5 years, an exceeding quantity of risk factors excluding smoking have been associated with the COPD development, predominantly in developing countries.

Exercise intolerance is a challenging result of COPD and often happens during arm activities. . Exercise intolerance can be best described by the concept of dynamic hyperinflation. The thoracic motion is regulated due to hyperinflation and thus capacity to increase tidal volume during exercise is limited. Many research studies have established that there is limited arm exercise capacity, and patients often complain of notable dyspnea and fatigue during arm activities essential in daily life. Two mechanisms have been recommended: neuro-mechanical dysfunction of respiratory musculature, that are diaphragm and accessory respiratory muscles, thoracic-abdominal asynchronous and changes in lung volume during upper limb activities. Impairments in ventilatory mechanics in COPD patients result in termination of arm exercises at lower workloads compared with healthy subjects.

When these patients were asked to open their mouths to breathe out instead of using pursed lips Breathing (PLB) they immediately developed severe dyspnea and suffocation. The term PLB was utilized as the patients had lips almost completely sealed while they were exhaling. However, the term pursed lip or puckered lip breathing was not well characterized, and the techniques taught to patients varied depending on the clinician. PLB was defined as a self-induced type of positive-pressure breath. One definition given by Wikipedia, is that PLB is a breathing technique that consists of exhaling through tightly pressed lip (pursed lips) and inhaling through nose with mouth closed. The "tightly" is the word that can be subjective and open to interpretation. The online free medical dictionary gives a very similar definition as Wikipedia; however, it removed "tightly" from the "tightly pursed lip". Regardless of "tightly pursed lip" vs. "pressed lip", the purpose of this breathing is to slow down the air flow during the exhalation to build up back pressure in the airway to avoid a sudden drop in intra-pulmonary pressure resulting in alveolar and airway collapse. Pursed lip breathing, is a strategic breathing training often used by COPD patients to obtain relief from dyspnea.

A shift in the pattern of recruitment of inspiratory and expiratory muscles with PLB exercise. There is a better activity in the rib cage and accessory muscles than with activity of diaphragm. The diaphragmatic tension-time index is decreased. Consequently, PLB by altering recruitment pattern decreases the possibility of fatigue of diaphragm and improves breathlessness. It also upsurges recruitment of abdominal expiratory musculature. Expiratory muscle recruitment does not only ease expiration but also aids in inspiration by developing the length-tension relationship of the inspiratory muscles.

Body positioning is one of the controlled breathing maneuvers to improve the respiratory muscle functioning and decreasing dyspnea. That is why the COPD patients often assume the tripod position, which is, sitting with forward lean of trunk and arm support, during breathlessness. This position develops the length-tension relationship of diaphragm and decreases the activity of sternocleidomastoid and scalene muscles thus improving thoraco-abdominal movement and reducing breathlessness. The arm support in this position recruits pectoralis major and pectoralis minor musculature to improve rib elevation

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate stage COPD according to GOLD criteria {i-e Global Initiative for Obstructive Lung Disease (GOLD) }

Exclusion Criteria:

* COPD patient with angina pectoris,
* third degree heart block,
* congestive heart failure and
* orthopedic or neuromuscular conditions (cervical involvement which aggravate symptoms) or radiculopathy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 1 week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 1 week
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters.
Peak Expiratory Flow (PEF) | 1 week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.
Oxygen Saturation (SpO2) | 1 week
  Changes from baseline SPO2 was measured in percentage. Oxygen immersion is the division of oxygen-soaked hemoglobin with respect to add up to hemoglobin in the blood. Pulse oximeter measure it.
Pulse Rate/Heart Rate | 1 week
  Changes from the Baseline, It is the speed of Pulse/heart contractions per minute. It is measured by pulse oximeter
Modified Borg Scale of Perceived Exertion | 1 week
  Changes from the Baseline, It is a subjective numeric scale ranging from 0 to 10, where 0 indicates "no dyspnea" and 10 indicates "unbearable dyspnea." A number is chosen by the patient in order to decide the best score that matches his level of dyspnea during physical activity.

SECONDARY OUTCOMES:
COPD Assessment Tool (CAT) | 1 week
  Changes from the baseline, CAT is a tool to assess the burden in COPD and is not a diagnostic tool. It is recommended by GOLD guidelines 2018. It is an eight item questionnaire with a scoring range of 0 to 40. It is categorized into four groups, that are, low(1) , medium(2), high(3) and very high(4) based on the level of effect of the disease on status of health. CAT has reliability of 0.85 to 0.98

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MsCPPT, Principal Investigator — Riphah International University
Locations (1):
- Department of Pulmonology of Rehman medical Institute., Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tunkamnerdthai O, Auvichayapat P, Punjaruk W, Manimmanakorn A, Leelayuwat N, Boonsawat W, et al. Modified Arm Swing Exercise Improves Oxidative Stress and Heart Rate Variability in Patients with Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Journal of Exercise Physiology Online. 2018;21(4)
- [Background] Halldin CN, Doney BC, Hnizdo E. Changes in prevalence of chronic obstructive pulmonary disease and asthma in the US population and associated risk factors. Chron Respir Dis. 2015 Feb;12(1):47-60. doi: 10.1177/1479972314562409. Epub 2014 Dec 24. PMID 25540134
- [Background] Ntritsos G, Franek J, Belbasis L, Christou MA, Markozannes G, Altman P, Fogel R, Sayre T, Ntzani EE, Evangelou E. Gender-specific estimates of COPD prevalence: a systematic review and meta-analysis. Int J Chron Obstruct Pulmon Dis. 2018 May 10;13:1507-1514. doi: 10.2147/COPD.S146390. eCollection 2018. PMID 29785100
- [Background] Mesquita Montes A, Maia J, Crasto C, de Melo CA, Carvalho P, Santos R, Pereira S, Vilas-Boas JP. Abdominal muscle activity during breathing in different postures in COPD "Stage 0" and healthy subjects. Respir Physiol Neurobiol. 2017 Apr;238:14-22. doi: 10.1016/j.resp.2017.01.001. Epub 2017 Jan 7. PMID 28082171
- [Background] Xu J, He S, Han Y, Pan J, Cao L. Effects of modified pulmonary rehabilitation on patients with moderate to severe chronic obstructive pulmonary disease: A randomized controlled trail. Int J Nurs Sci. 2017 Jun 27;4(3):219-224. doi: 10.1016/j.ijnss.2017.06.011. eCollection 2017 Jul 10. PMID 31406744
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Bharadwaj TA, Jiandani MP, Mehta A. PURSED LIP BREATHING INCREASES UNSUPPORTED UPPER EXTREMITY EXERCISE ENDURANCE AND REDUCES DESATURATION IN COPD. Romanian Journal of Physical Therapy/Revista Romana de Kinetoterapie. 2016;21(38).